CLINICAL TRIAL: NCT06137833
Title: Clinical Study on Wide Spectrum Micronutrients Supplementation in Patients With Cancer Related Fatigue During Neoadjuvant and Adjuvant Chemotherapy
Brief Title: Wide Spectrum Micronutrients Supplementation in Patients With Cancer Related Fatigue During Neoadjuvant and Adjuvant Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanutra S.p.a. (Industry)
Collaborators: Latis S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: APPORTAL-01-23
Record Dates: First submitted 2023-07-16; First posted 2023-11-18 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Fatigue; Breast Cancer
MeSH Terms: conditions — Fatigue; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- APPORTAL® (Experimental): APPORTAL® sachet, 1 sachet per day dissolved in a glass of water. To be consumed in the morning, about 10 minutes after breakfast. Dosage form: powder Route: Oral Treatment duration: 8 weeks
  Interventions: Dietary Supplement: APPOPRTAL®
- PLACEBO (Placebo Comparator): PLACEBO sachet, 1 sachet per day dissolved in a glass of water To be consumed in the morning, about 10 minutes after breakfast. Dosage form: powder Route: Oral Treatment duration: 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: APPOPRTAL® — 1 sachet of APPORTAL® contains: Vitamin C 37,5 mg; Vitamin E 30 mg; Vitamin PP 18 mg; Vitamin B1 1 mg; Vitamin D 25 μg; Vitamin H 25 μg; L-arginine 1000 mg; L-carnitine 500 mg; Taurine 25 mg; Ginseng e.s. 100 mg; Eleutherococcus e.s. 50 mg; Magnesium 187,5 mg; Iron 14 mg; Zinc 1,5 mg; Iodine 75 μg; Selenium 27,5 μg; Coenzyme Q10 100 mg; Lycopene 3,06 mg; Tocotrienols 2,5 mg; Coenzyme Q10 100 mg; Lycopene 3,06 mg; Tocotrienols 2,5 mg
  Arms: APPORTAL®
Other: Placebo — Ingredients: Maltodextrin, acidifying agent: citric acid, flavours, anticaking agent: tricalcium phosphate, beetroot juice powder; sweetener: sucralose, anti-caking agent: silicon dioxide, colouring agent: beta-carotene
  Arms: PLACEBO

SUMMARY:
The goal of this clinical trial is to test the effect of the administration of APPORTAL® in addition to the SoC (recommended physical exercise), in patients with breast cancer, suffering from fatigue during neoadjuvant and adjuvant chemotherapy. The main questions it aims to answer are:

* if the food supplement APPORTAL® can be of help in supporting the physiological energy level, against the fatigue symptom in cancer patients undergoing adjuvant chemotherapy;
* if the supplementation with APPORTAL® can optimize the nutritional status, the muscular strength, the quality of life of the patient.

Also, the patients' satisfaction on the product received, the adherence to treatment will be evaluated and the overall safety and tolerability of the study product.

The patients will be asked to perform 3 study visits from baseline to the end of treatment (at 4 and 8 weeks after baseline) and a follow-up visit after 12 weeks from baseline.

The main assessments at each visit will be:

* physical examination, weight, Body Mass Index (BMI), body temperature (°C), heart rate, respiratory frequency, and systolic and diastolic blood pressure;
* previous and concomitant treatments;
* fatigue assessment through BFI questionnaire;
* quality of life through questionnaire SF-12;
* muscular strength (dynamometer)
* Adverse Event check (from Visit 2) Moreover, at visit 1 (baseline) and at visit 3 (end of treatment) a blood sample will be collected to evaluate the blood metabolites.

Telephonic follow-up will be done at 2 weeks, 6 weeks, 10 weeks to assess compliance and to recommendations on physical activity and to study treatment (only at 2 and 6 weeks) and tolerability/safety.

Participants will receive the nutrition supplement or the placebo, in addition to the SoC (recommended physical exercise), for 8 weeks.

Researchers will compare Apportal® and Placebo groups to see if the physiological energy level against the fatigue symptom, the nutritional status, the muscular strength, the quality of life of the patient improve after 8 weeks of treatment with APPORTAL® in addition to SoC (recommended physical exercise).

DETAILED DESCRIPTION:
SAMPLE SIZE DETERMINATION Considering the average of the BFI 5 in the placebo group and the average 3 in the treated group, with standard deviation of 3, power at 80% and alpha 0.05, we obtain 37 patients per group, thus a total of 74 patients. If a drop-out rate of 20% is fixed, 92 patients in total are obtained. So, a sample of 92 subjects would be sufficient.

DATA SAFETY MONITORING BOARD / DATA MONITORING COMMITTEE No Data Safety Monitoring Board (DSMB) or Data Monitoring Committee (DMC) will be convened for the evaluation of safety data during the study. However, the Network Italiano Cure di Supporto in Oncologia (NICSO) society will be in charge of the evaluation of safety information. In fact, a Scientific Committee, composed by NICSO members, has been established to support the Sponsor in the continuous evaluation of safety data emerging from the study.

MONITORING AND QUALITY ASSURANCE The study will be monitored by adequately qualified and trained clinical monitors. Before the start of the study, the CRO (Contract Research Organization) responsible for the study site has the task to assess the adequacy of the study site and the staff involved. After start, the study will be monitored to ensure the proper conduct of the clinical study.

DATA COLLECTION An Electronic Case Report Form (e-CRF) will be used for recording patient's study data.

The Investigator will maintain a list of all persons authorized to make entries and/or corrections on the CRFs. Each authorized person will be provided with a user-specific ID (Identification) protected by a renewable password. Data entries and corrections will be made only by the authorized persons. The e-CRF system will record date and time of any entry and /or correction and the user ID of the person making the entry/correction. The system will keep track of all old and new values (audit trail).

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 18 or higher.
2. Patients diagnosed with histologically confirmed breast cancer.
3. Patients having done at least one cycle of neoadjuvant or adjuvant chemotherapy (independently from type of chemotherapy) and who are on active chemotherapy treatment throughout the duration of the study (*).
4. Patients with ECOG performance status ≤1 at screening.
5. Patients with cancer related fatigue of moderate-severe intensity (Numerical Rating Scale NRS > 4).
6. Patients able to follow the recommendations on the physical exercise to do.
7. Patients who accept to use adequate contraceptive methods, if they are of child-bearing potential.
8. Patients willing and able to give signed informed consent and, in the opinion of the Investigator, to comply with the protocol tests and procedures.

(*)Examples of chemotheraphy and standard therapeutic regimens in the neoadjuvant and adjuvant phase in breast cancer and on the basis of the biological characteristics of the neoplasm are as follows:

Neoadjuvant Chemotheraphy

* Epirubicin + Cyclophosphamide, 3 cycles -> Taxol* weekly for 12 weeks;
* Epirubicin + Cyclophosphamide -> Pertuzumab + Trastuzumab (or Phesgo) 3 cycles + Taxol weekly for 12 weeks;
* Carboplatin + Taxol* weekly for 12 weeks -> Epirubicin + Cyclophosphamide;

  * Taxol could be replaced by Taxotere

Adjuvant Chemotheraphy

* Epirubicin + Cyclophosphamide, 4 cycles, every 21 days -> Taxol weekly for 12 weeks
* Epirubicin + Cyclophosphamide, 4 cycles, every 14 days -> Taxol, 4 cycles every 14 days
* Epirubicin + Cyclophosphamide, 4 cycles every 21 days -> Taxol weekly + Trastuzumab with or without Pertuzumab for 1 year
* Taxotere + Cyclophosphamide, 4 cycles, every 21 days.

These lists are not to be considered exclusive

Exclusion Criteria:

1. Women who are pregnant or breast-feeding.
2. Neoplastic disease other than primary breast cancer.
3. Had major surgery other than breast cancer surgery (central venous access placement and tumor biopsies are not considered major surgery) within 4 weeks prior to randomization. Patients must be well recovered from acute effects of surgery prior to screening. Patients should not have plans to undergo major surgical procedures during the treatment period.
4. Patients with known or symptomatic metastases.
5. Patients unable to readily swallow. Patients with severe gastrointestinal disease (including esophagitis, gastritis, malabsorption, or obstructive symptoms) or intractable or frequent vomiting are excluded.
6. Patients with known or suspected allergy or hypersensitivity to the study products or any of their excipients.
7. Patients with an active, uncontrolled infection.
8. Patients with uncontrolled diabetes mellitus.
9. Patients with untreated clinically relevant hypothyroidism.
10. Patients with concomitant not-correctable alterations, present before chemotherapy, possible determinants of fatigue (NRS ≥ 4), such as anemia, not well controlled pain (NRS > 4), insomnia, electrolyte imbalance, dehydration, anorexia/cachexia, hepatic, renal or heart failure, adrenocortical failure, neurological deficit.
11. Other clinical diagnosis, serious chronic diseases (renal failure with creatinine clearance <30 ml / min; liver failure, heart failure with NYHA -New York Heart Association- class> 2), ongoing or intercurrent illness that in the Investigator's opinion would prevent the patient's participation.
12. Patients receiving opioids or corticosteroids (except as replacement therapy at physiological dose, in subjects with adrenal insufficiency or to prevent emesis on the chemotherapy day).
13. Patients receiving parenteral nutrition (either total or partial).
14. Use of other investigational drug(s) within 30 days before study entry or during the study.
15. Triple negative patients in neoadjuvant treatment with Pembrolizumab.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of fatigue perception by the patient through the BFI questionnaire | Change from baseline to 8 weeks of treatment (Visit 3), in active and placebo groups.
  The Brief Fatigue Inventory (BFI) is a questionnaire specifically developed for rapid assessment of CRF. It is a simple, easily administered questionnaire and the fatigue scale (validated in different languages) consists in nine items anticipated by a flag question asking the patient whether she has felt unusually fatigued or tired during the last week. Three items are related to the intensity of fatigue "right now", at its "usual" level and at its "worst" level during the past 24 h using a 0-10 numerical scale (0= no fatigue, 10= fatigue as bad as you can image). Six items measure the interference of fatigue with the patients' life during the past 24 h by a 0-10 numerical scale (0= does not interfere, 10= completely interferes). Higher scores represent to more severe fatigue

SECONDARY OUTCOMES:
The change of fatigue perception by the patient through the BFI questionnaire | Change after 4, 8 and 12 weeks with respect to baseline in both the active and placebo groups
  The Brief Fatigue Inventory (BFI) is a questionnaire specifically developed for rapid assessment of CRF. It is a simple, easily administered questionnaire and the fatigue scale (validated in different languages) consists in nine items anticipated by a flag question asking the patient whether she has felt unusually fatigued or tired during the last week. Three items are related to the intensity of fatigue "right now", at its "usual" level and at its "worst" level during the past 24 h using a 0-10 numerical scale (0= no fatigue, 10= fatigue as bad as you can image). Six items measure the interference of fatigue with the patients' life during the past 24 h by a 0-10 numerical scale (0= does not interfere, 10= completely interferes). Higher scores represent to more severe fatigue
Change in Iron status through hemoglobin assessment | Change after 8 weeks of study treatment with respect to baseline, in both the active and placebo groups
  Blood samples of about 5 mL will be collected for the assessment of iron status (hemoglobin, ferritin, transferrin saturation), nutritional markers (albumin, total cholesterol, HDL, LDL and triglycerides), oxidative markers (homocysteine, uric acid) and C-Reactive Protein, serum L-arginine levels. Blood samples will be analysed locally by each site laboratory.
Change in Iron status through ferritin assessment | Change after 8 weeks of study treatment with respect to baseline, in both the active and placebo groups
  Blood samples of about 5 mL will be collected for the assessment of iron status (hemoglobin, ferritin, transferrin saturation), nutritional markers (albumin, total cholesterol, HDL, LDL and triglycerides), oxidative markers (homocysteine, uric acid) and C-Reactive Protein, serum L-arginine levels. Blood samples will be analysed locally by each site laboratory.
Change in Iron status through transferrin saturation assessment | Change after 8 weeks of study treatment with respect to baseline in both the active and placebo groups
  Blood samples of about 5 mL will be collected for the assessment of iron status (hemoglobin, ferritin, transferrin saturation), nutritional markers (albumin, total cholesterol, HDL, LDL and triglycerides), oxidative markers (homocysteine, uric acid) and C-Reactive Protein, serum L-arginine levels. Blood samples will be analysed locally by each site laboratory.
Change in nutritional status through albumin assessment | Change after 8 weeks of study treatment with respect to baseline in both the active and placebo groups
  Blood samples of about 5 mL will be collected for the assessment of iron status (hemoglobin, ferritin, transferrin saturation), nutritional markers (albumin, total cholesterol, HDL, LDL and triglycerides), oxidative markers (homocysteine, uric acid) and C-Reactive Protein, serum L-arginine levels. Blood samples will be analysed locally by each site laboratory.
Change in nutritional status through assessment of total cholesterol, HDL, LDL and triglycerides | Change after 8 weeks of study treatment with respect to baseline in both the active and placebo groups
  Blood samples of about 5 mL will be collected for the assessment of iron status (hemoglobin, ferritin, transferrin saturation), nutritional markers (albumin, total cholesterol, HDL, LDL and triglycerides), oxidative markers (homocysteine, uric acid) and C-Reactive Protein, serum L-arginine levels. Blood samples will be analysed locally by each site laboratory.
Change in oxidative status through homocysteine assessment | Change after 8 weeks of study treatment with respect to baseline in both the active and placebo groups
  Blood samples of about 5 mL will be collected for the assessment of iron status (hemoglobin, ferritin, transferrin saturation), nutritional markers (albumin, total cholesterol, HDL, LDL and triglycerides), oxidative markers (homocysteine, uric acid) and C-Reactive Protein, serum L-arginine levels. Blood samples will be analysed locally by each site laboratory.
Change in oxidative status through uric acid assessment | Change after 8 weeks of study treatment with respect to baseline in both the active and placebo groups
  Blood samples of about 5 mL will be collected for the assessment of iron status (hemoglobin, ferritin, transferrin saturation), nutritional markers (albumin, total cholesterol, HDL, LDL and triglycerides), oxidative markers (homocysteine, uric acid) and C-Reactive Protein, serum L-arginine levels. Blood samples will be analysed locally by each site laboratory.
Change in oxidative status through C-Reactive Protein (CRP) assessment | Change after 8 weeks of study treatment with respect to baseline in CRP in both the active and placebo groups
  Blood samples of about 5 mL will be collected for the assessment of iron status (hemoglobin, ferritin, transferrin saturation), nutritional markers (albumin, total cholesterol, HDL, LDL and triglycerides), oxidative markers (homocysteine, uric acid) and C-Reactive Protein, serum L-arginine levels. Blood samples will be analysed locally by each site laboratory.
Change in serum L-arginina levels | Change after 8 weeks of study treatment with respect to baseline in both the active and placebo groups
  Blood samples of about 5 mL will be collected for the assessment of iron status (hemoglobin, ferritin, transferrin saturation), nutritional markers (albumin, total cholesterol, HDL, LDL and triglycerides), oxidative markers (homocysteine, uric acid) and C-Reactive Protein, serum L-arginine levels. Blood samples will be analysed locally by each site laboratory.
Changes in QoL through SF-12 Questionnaire | Change after 4, 8 and 12 weeks with respect to baseline in both the active and placebo groups
  SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
  The SF-12 is a shortened version of it's predecessor, the SF-36 and it was created to reduce the burden of response The SF-12 consists of twelve questions that measure the same eight domains as the SF-36, to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). Mental health-related scales include Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH).
Change in muscular strength (hand grip test), | Change after 4, 8 and 12 weeks with respect to baseline in both the active and placebo groups
  Grip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles. It can be used as a screening tool for the measurement of upper body strength and overall strength. Within this clinical study an hand digital dynamometer will be used.
Overall patient's satisfaction with the product received, through a 5-points Likert scale | End of treatment (after 8 weeks of study treatment), in both the active and placebo groups
  5-points Likert scale: 1=very satisfied, 2=satisfied, 3=not satisfied nor unsatisfied, 4=not satisfied, 5= not satisfied at all
Adherence to treatment | After 4 weeks and after 8 weeks from baseline
  The percentage of actual sachets taken by the patient in relation to the expected number of sachets, calculated as (number of real sachets taken / number of expected sachets) * 100

OTHER OUTCOMES:
Study product tolerability | Through study completion, an average of 12 weeks, in active and placebo groups
  Study product tolerability will be assessed by number of adverse events related to the product
Change in Physical Examination through weight measurement | Change after 4, 8 and 12 weeks from baseline in both the active and placebo groups
  Weight (Kg)
Change in Physical Examination through BMI evaluation | Change after 4, 8 and 12 weeks from baseline in both the active and placebo groups
  BMI (Kg/m^2)
Change in Physical Examinations through clinical evaluation by system | After 4, 8 and 12 weeks from baseline in both the active and placebo groups
  Number of normal/abnormal conditions per system
Change in vital signs through body temperature measurement | Change after 4, 8 and 12 weeks from baseline in Body temperature, in both the active and placebo groups
  Body temperature °C
Change in vital signs through Respiratory Frequency measurement | Change after 4, 8 and 12 weeks from baseline in Heart Rate, in both the active and placebo groups
  Respiratory Frequency (rpm)
Change in vital signs through Heart Rate measurement | Change after 4, 8 and 12 weeks from baseline in both the active and placebo groups
  Heart Rate (bpm)
Change in vital signs through blood pressure measurement | Change after 4, 8 and 12 weeks from baseline in both the active and placebo groups
  Systolic and Diastolic blood pressure (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Fabi, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (5):
- Italy (5):
  - U.O.C. Oncologia medica ASST Spedali Civili di Brescia, Brescia, BRESCIA
  - Cancer Center U.O. Oncologia Medica ed Ematologia IRCCS Humanitas Research Hospital, Rozzano, MILANO
  - U.O. Oncologia 2 Universitaria A.O.U. Pisana, Pisa, PISA
  - UOSD di Medicina di Precisione e Senologia, Policlinico Universitario A. Gemelli, Rome, ROME
  - Dipartimento di Oncologia Azienda Sanitaria Universitaria Integrata di Udine, Udine, UDINE

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Jemal A, Center MM, DeSantis C, Ward EM. Global patterns of cancer incidence and mortality rates and trends. Cancer Epidemiol Biomarkers Prev. 2010 Aug;19(8):1893-907. doi: 10.1158/1055-9965.EPI-10-0437. Epub 2010 Jul 20. PMID 20647400
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2012. CA Cancer J Clin. 2012 Jan-Feb;62(1):10-29. doi: 10.3322/caac.20138. Epub 2012 Jan 4. PMID 22237781
- [Background] Mortimer JE, Barsevick AM, Bennett CL, Berger AM, Cleeland C, DeVader SR, Escalante C, Gilreath J, Hurria A, Mendoza TR, Rugo HS. Studying cancer-related fatigue: report of the NCCN scientific research committee. J Natl Compr Canc Netw. 2010 Dec;8(12):1331-9. doi: 10.6004/jnccn.2010.0101. PMID 21147900
- [Background] Ruiz-Casado A, Alvarez-Bustos A, de Pedro CG, Mendez-Otero M, Romero-Elias M. Cancer-related Fatigue in Breast Cancer Survivors: A Review. Clin Breast Cancer. 2021 Feb;21(1):10-25. doi: 10.1016/j.clbc.2020.07.011. Epub 2020 Jul 24. PMID 32819836
- [Background] So WK, Marsh G, Ling WM, Leung FY, Lo JC, Yeung M, Li GK. The symptom cluster of fatigue, pain, anxiety, and depression and the effect on the quality of life of women receiving treatment for breast cancer: a multicenter study. Oncol Nurs Forum. 2009 Jul;36(4):E205-14. doi: 10.1188/09.ONF.E205-E214. PMID 19581224
- [Background] Gaston-Johansson F, Fall-Dickson JM, Bakos AB, Kennedy MJ. Fatigue, pain, and depression in pre-autotransplant breast cancer patients. Cancer Pract. 1999 Sep-Oct;7(5):240-7. doi: 10.1046/j.1523-5394.1999.75008.x. PMID 10687593
- [Background] Berger AM, Abernethy AP, Atkinson A, Barsevick AM, Breitbart WS, Cella D, Cimprich B, Cleeland C, Eisenberger MA, Escalante CP, Jacobsen PB, Kaldor P, Ligibel JA, Murphy BA, O'Connor T, Pirl WF, Rodler E, Rugo HS, Thomas J, Wagner LI. NCCN Clinical Practice Guidelines Cancer-related fatigue. J Natl Compr Canc Netw. 2010 Aug;8(8):904-31. doi: 10.6004/jnccn.2010.0067. No abstract available. PMID 20870636
- [Background] Cella D, Davis K, Breitbart W, Curt G; Fatigue Coalition. Cancer-related fatigue: prevalence of proposed diagnostic criteria in a United States sample of cancer survivors. J Clin Oncol. 2001 Jul 15;19(14):3385-91. doi: 10.1200/JCO.2001.19.14.3385. PMID 11454886
- [Background] Sadler IJ, Jacobsen PB, Booth-Jones M, Belanger H, Weitzner MA, Fields KK. Preliminary evaluation of a clinical syndrome approach to assessing cancer-related fatigue. J Pain Symptom Manage. 2002 May;23(5):406-16. doi: 10.1016/s0885-3924(02)00388-3. PMID 12007758
- [Background] Mustian KM, Alfano CM, Heckler C, Kleckner AS, Kleckner IR, Leach CR, Mohr D, Palesh OG, Peppone LJ, Piper BF, Scarpato J, Smith T, Sprod LK, Miller SM. Comparison of Pharmaceutical, Psychological, and Exercise Treatments for Cancer-Related Fatigue: A Meta-analysis. JAMA Oncol. 2017 Jul 1;3(7):961-968. doi: 10.1001/jamaoncol.2016.6914. PMID 28253393
- [Background] Puetz TW, Herring MP. Differential effects of exercise on cancer-related fatigue during and following treatment: a meta-analysis. Am J Prev Med. 2012 Aug;43(2):e1-24. doi: 10.1016/j.amepre.2012.04.027. PMID 22813691
- [Background] Mishra SI, Scherer RW, Geigle PM, Berlanstein DR, Topaloglu O, Gotay CC, Snyder C. Exercise interventions on health-related quality of life for cancer survivors. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD007566. doi: 10.1002/14651858.CD007566.pub2. PMID 22895961
- [Background] Fabi A, Bhargava R, Fatigoni S, Guglielmo M, Horneber M, Roila F, Weis J, Jordan K, Ripamonti CI; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Cancer-related fatigue: ESMO Clinical Practice Guidelines for diagnosis and treatment. Ann Oncol. 2020 Jun;31(6):713-723. doi: 10.1016/j.annonc.2020.02.016. Epub 2020 Mar 12. No abstract available. PMID 32173483
- [Background] Horneber M, Bueschel G, Dennert G, Less D, Ritter E, Zwahlen M. How many cancer patients use complementary and alternative medicine: a systematic review and metaanalysis. Integr Cancer Ther. 2012 Sep;11(3):187-203. doi: 10.1177/1534735411423920. Epub 2011 Oct 21. PMID 22019489
- [Background] Boon HS, Olatunde F, Zick SM. Trends in complementary/alternative medicine use by breast cancer survivors: comparing survey data from 1998 and 2005. BMC Womens Health. 2007 Mar 30;7:4. doi: 10.1186/1472-6874-7-4. PMID 17397542
- [Background] Greenlee H, Kwan ML, Ergas IJ, Strizich G, Roh JM, Wilson AT, Lee M, Sherman KJ, Ambrosone CB, Hershman DL, Neugut AI, Kushi LH. Changes in vitamin and mineral supplement use after breast cancer diagnosis in the Pathways Study: a prospective cohort study. BMC Cancer. 2014 May 29;14:382. doi: 10.1186/1471-2407-14-382. PMID 24884705
- [Background] Greenlee H, Kwan ML, Ergas IJ, Sherman KJ, Krathwohl SE, Bonnell C, Lee MM, Kushi LH. Complementary and alternative therapy use before and after breast cancer diagnosis: the Pathways Study. Breast Cancer Res Treat. 2009 Oct;117(3):653-65. doi: 10.1007/s10549-009-0315-3. Epub 2009 Jan 31. PMID 19184414
- [Background] Link AR, Gammon MD, Jacobson JS, Abrahamson P, Bradshaw PT, Terry MB, Teitelbaum S, Neugut A, Greenlee H. Use of Self-Care and Practitioner-Based Forms of Complementary and Alternative Medicine before and after a Diagnosis of Breast Cancer. Evid Based Complement Alternat Med. 2013;2013:301549. doi: 10.1155/2013/301549. Epub 2013 Aug 12. PMID 23997792
- [Background] Matsuno RK, Pagano IS, Maskarinec G, Issell BF, Gotay CC. Complementary and alternative medicine use and breast cancer prognosis: a pooled analysis of four population-based studies of breast cancer survivors. J Womens Health (Larchmt). 2012 Dec;21(12):1252-8. doi: 10.1089/jwh.2012.3698. Epub 2012 Oct 17. PMID 23075455
- [Background] Bright-Gbebry M, Makambi KH, Rohan JP, Llanos AA, Rosenberg L, Palmer JR, Adams-Campbell LL. Use of multivitamins, folic acid and herbal supplements among breast cancer survivors: the black women's health study. BMC Complement Altern Med. 2011 Apr 15;11:30. doi: 10.1186/1472-6882-11-30. PMID 21496245
- [Background] Rossato MS, Brilli E, Ferri N, Giordano G, Tarantino G. Observational study on the benefit of a nutritional supplement, supporting immune function and energy metabolism, on chronic fatigue associated with the SARS-CoV-2 post-infection progress. Clin Nutr ESPEN. 2021 Dec;46:510-518. doi: 10.1016/j.clnesp.2021.08.031. Epub 2021 Sep 6. PMID 34857243
- [Background] Galluzzo V, Zazzara MB, Ciciarello F, Savera G, Pais C, Calvani R, Picca A, Marzetti E, Landi F, Tosato M; Gemelli Against COVID-19 Post-Acute Care Team. Fatigue in Covid-19 survivors: The potential impact of a nutritional supplement on muscle strength and function. Clin Nutr ESPEN. 2022 Oct;51:215-221. doi: 10.1016/j.clnesp.2022.08.029. Epub 2022 Aug 31. PMID 36184207
- [Background] Cho J, Park W, Lee S, Ahn W, Lee Y. Ginsenoside-Rb1 from Panax ginseng C.A. Meyer activates estrogen receptor-alpha and -beta, independent of ligand binding. J Clin Endocrinol Metab. 2004 Jul;89(7):3510-5. doi: 10.1210/jc.2003-031823. PMID 15240639
- [Background] Hao K, Gong P, Sun SQ, Hao HP, Wang GJ, Dai Y, Liang Y, Xie L, Li FY. Beneficial estrogen-like effects of ginsenoside Rb1, an active component of Panax ginseng, on neural 5-HT disposition and behavioral tasks in ovariectomized mice. Eur J Pharmacol. 2011 May 20;659(1):15-25. doi: 10.1016/j.ejphar.2011.03.005. Epub 2011 Mar 22. PMID 21414307
- [Background] Fan M, Shan M, Lan X, Fang X, Song D, Luo H, Wu D. Anti-cancer effect and potential microRNAs targets of ginsenosides against breast cancer. Front Pharmacol. 2022 Oct 5;13:1033017. doi: 10.3389/fphar.2022.1033017. eCollection 2022. PMID 36278171
- [Background] Malati CY, Robertson SM, Hunt JD, Chairez C, Alfaro RM, Kovacs JA, Penzak SR. Influence of Panax ginseng on cytochrome P450 (CYP)3A and P-glycoprotein (P-gp) activity in healthy participants. J Clin Pharmacol. 2012 Jun;52(6):932-9. doi: 10.1177/0091270011407194. Epub 2011 Jun 6. PMID 21646440
- [Background] Mendoza TR, Wang XS, Cleeland CS, Morrissey M, Johnson BA, Wendt JK, Huber SL. The rapid assessment of fatigue severity in cancer patients: use of the Brief Fatigue Inventory. Cancer. 1999 Mar 1;85(5):1186-96. doi: 10.1002/(sici)1097-0142(19990301)85:53.0.co;2-n. PMID 10091805
- [Background] Catania G, Bell C, Ottonelli S, Marchetti M, Bryce J, Grossi A, Costantini M. Cancer-related fatigue in Italian cancer patients: validation of the Italian version of the Brief Fatigue Inventory (BFI). Support Care Cancer. 2013 Feb;21(2):413-9. doi: 10.1007/s00520-012-1539-z. Epub 2012 Jul 13. PMID 22790224
- See also: American Cancer Society. Cancer facts & figures 2012 — https://www.cancer.org/research/cancer-facts-statistics/all-cancer-facts-figures/cancer-facts-figures-2012.html
- See also: 12-Item Short Form Survey (SF-12) - Standard Italian Version — https://www.studocu.com/it/document/universita-degli-studi-di-torino/psiconcologia-e-cure-palliative-psycho-oncology/sf12-questionario/11590607